CLINICAL TRIAL: NCT00097149
Title: Systematic Pediatric Care for Oral Clefts - South America
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of Iowa (Other); Latin-American Collaborative Study of Congenital Malformations (ECLAMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN 04 Aim II; U01HD040561 (NIH)
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Cleft Lip; Cleft Palate; Congenital Defects
Keywords: Congenital birth defects; Cleft lip; Cleft palate; Global Network; Neurodevelopmental outcome; Maternal and child health; International; Women's health; Brazil; Brasil; Latin America; ECLAMC; Argentina; Bolivia; Chile; Colombia; Ecuador; Venezuela
MeSH Terms: conditions — Cleft Lip; Cleft Palate; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Systematic pediatric care

SUMMARY:
Cleft lip and palate are a significant component of morbid human birth defects in the developing world. This study measures the impact of having a child born with a cleft lip on subsequent maternal/infant family health, and whether frequent pediatric care compared to standard pediatric care will reduce neonatal mortality in children born with cleft lip and palate.

DETAILED DESCRIPTION:
Craniofacial anomalies and cleft lip with or without cleft palate (CL/P) are a model for the impact of birth defects on fetal and neonatal health directly and maternal health indirectly. Craniofacial anomalies comprise a significant component of morbid human birth defects. This study is composed of two Subprojects, A and B. Subproject A involves provision of intensive pediatric care over the first 28 days of life for a prospective group of about 694 cleft cases, which will be compared to a retrospective group of about 464 cleft cases. Nonsyndromic cleft lip with or without cleft palate (NSCL/P) cases (about 264 cases) of Subproject A will be randomized into two groups: intervened (about 132 cases) and non-intervened (about 132 cases). Sub-project B involves provision of systematic pediatric care over a 2-year period for the intervened group. This group will be compared to the non-intervened group in order to study the effect of the intervention on the neurodevelopment and physical health of the child as well as the emotional and social health of the family. The standard care group also will be compared to a group of about 264 healthy controls, matched by sex and place and date of birth in order to study the impact of the cleft on the physical health and neurodevelopment of the child as well as the emotional and social health of the family. The importance of the study relates to the substantial burden caused by clefts and the necessity of developing and testing approaches that may lessen this burden. The outcomes of this project will be to further strengthen collaborative relationships in the area of craniofacial anomalies between South America and the United States; to better understand the effects of birth defects, and craniofacial anomalies in particular, on maternal family units; and, to decrease the burden of these defects directly. The sample size was based on an expected overall 28 days mortality rate among cleft infants that is around 0.25, calculated at a 0.05 significance level.

ELIGIBILITY:
Subproject A:

* All children born with an oral cleft in a participating hospital (hospitals in Argentina, Bolivia, Brazil, Chile, Colombia and Venezuela affiliated with ECLAMC)

Subproject B: Cases from Subproject A that meet the following criteria:

* Cleft lip with or without cleft palate or cleft palate only
* Birth weight >2500 g
* No other identifiable birth defect: nonsyndromic
* Singleton (nonmultiple birth)
* No other complications requiring systematic care

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 696
Dates: Start 2003-05; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
SUBPROJECT A: Neonatal mortality
SUBPROJECT B: Neurodevelopmental outcome
Weight

SECONDARY OUTCOMES:
SUBPROJECT A: Hospitalizations, Weight
SUBPROJECT B: Height, Speech, Hearing, Mortality, Cleft surgery, Rate of weight gain, Financial burden, Syndromic classification, Emotional and social family development

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Murray, M.D., Principal Investigator — University of Iowa
Locations (1):
- Latin-American Collaborative Study of Congenital Malformations (ECLAMC), Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Wehby GL, Castilla EE, Goco N, Rittler M, Cosentino V, Javois L, Kindem M, Chakraborty H, Dutra G, Lopez-Camelo JS, Orioli IM, Murray JC. The effect of systematic pediatric care on neonatal mortality and hospitalizations of infants born with oral clefts. BMC Pediatr. 2011 Dec 28;11:121. doi: 10.1186/1471-2431-11-121. PMID 22204448
- [Derived] Wehby GL, Castilla EE, Goco N, Rittler M, Cosentino V, Javois L, McCarthy AM, Bobashev G, Litavecz S, Mariona A, Dutra G, Lopez-Camelo JS, Orioli IM, Murray JC. Description of the methodology used in an ongoing pediatric care interventional study of children born with cleft lip and palate in South America [NCT00097149]. BMC Pediatr. 2006 Mar 24;6:9. doi: 10.1186/1471-2431-6-9. PMID 16563165
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: RTI International — http://www.rti.org/